CLINICAL TRIAL: NCT02866734
Title: The Feasibility of Screening for Diabetic Retinopathy in Private Practice Hong Kong
Brief Title: Diabetic Retinopathy Screening in Private Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12133951
Record Dates: First submitted 2016-07-27; First posted 2016-08-15 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Retinopathy; Screening; Fee for screening; Private practice
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Free screening group (Active Comparator): Subjects in this group receive free diabetic retinopathy screening.
  Interventions: Other: Free screening group
- Pay screening group ($150) (Active Comparator): Subjects in this group receiving diabetic retinopathy screening will be charged HK$150.
  Interventions: Other: Pay screening group ($150)
- Pay screening group ($300) (Active Comparator): Subjects in this group receiving diabetic retinopathy screening will be charged HK$300.
  Interventions: Other: Pay screening group ($300)

INTERVENTIONS:
Other: Free screening group — The intervention provide Diabetic Retinopathy screening without charging a fee.
  Arms: Free screening group
Other: Pay screening group ($150) — The intervention is charging HK$150 for the Diabetic Retinopathy screening.
  Arms: Pay screening group ($150)
Other: Pay screening group ($300) — The intervention is charging HK$300 for the Diabetic Retinopathy screening.
  Arms: Pay screening group ($300)

SUMMARY:
Introduction: Diabetic mellitus (DM) is a prevalent disease in Hong Kong (HK) and diabetic retinopathy (DR) is one of the most common complications of DM. Screening for DR is a cost-effective method to identify patients who are at risk of vision loss so that timely treatment can be provided to patients. In Hong Kong, the Hospital Authority has recently set up screening services (RAMP) in the government outpatient clinics and all DM patients attending these clinics will be screened at least once every two years and some every six months, according to their individual risks. However, those diabetic patients who attend the private sector for their primary care may not have access to this service.

Aim: This study from the University of Hong Kong aims to determine the characteristics of a sustainable approach to setting up an effective and quality-controlled screening service for DR in the private primary care sector of Hong Kong and to estimate the potential benefit to be gained in terms of impact on avoidable vision loss, costs of care and potential for further development of this model in chronic disease care.

Methods:A screening centre is being set up and a randomised study carried out in which screening will be offered at three different fee levels to subjects recruited by their general practitioner (GP). The following data will be collected (a) willingness to attend screening at the different fee levels (b) screening findings in terms of DR and other eye diseases (c) risk factors and other characteristics of those screened and unscreened. The information will allow us to estimate the level of fee which best combines effectiveness with sustainability in the longer term.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed to have diabetic mellitus
* Able to give informed consent

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
The overall, & at different fee level, uptake (as a percentage of participants) of screening from those at-risk patients who attend private GP's | one year

SECONDARY OUTCOMES:
Percentage of participants with diabetes who are only under the care of a private GP, or also attend specialist service, and have had access to DR screening | one year
Prevalence of DR (overall, and for sight-threatening diabetic retinopathy) among diabetic patients in private primary care | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Cheuk Hung Chan, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Ophthalmology, The University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No